CLINICAL TRIAL: NCT00882817
Title: Effects of Pulmonary Rehabilitation in Interstitial Lung Diseases: a Prospective Randomized Controlled Trial
Brief Title: Pulmonary Rehabilitation in Interstitial Lung Diseases
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Marc Decramer, Prof. Dr., KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B32220095560; S1490
Record Dates: First submitted 2009-04-15; First posted 2009-04-17 (Estimated); Last update posted 2013-08-01 (Estimated); Status verified 2013-07

CONDITIONS: Interstitial Lung Disease
Keywords: ILD
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Pulmonary Rehabilitation
  Interventions: Other: Pulmonary Rehabilitation
- 2 (No Intervention)

INTERVENTIONS:
Other: Pulmonary Rehabilitation — The intervention group will perform a 6 month pulmonary rehabilitation program which consists of training, patient education, nutrition counseling and psychosocial support. They will be evaluated with some tests for the study.
  Arms: 1

SUMMARY:
Treatment in interstitial lung diseases (ILD) is frequently ineffective. Pulmonary rehabilitation (PR) is an excellent therapeutic option in another chronic lung diseases such as chronic obstructive pulmonary disease (COPD). This prospective randomized controlled study aims to evaluate the short and long-term effects of PR in patients with ILD. For this purpose, 60 ILD patients will be randomly assigned to a PR or a control group.

The investigators hypothesize that PR will improve exercise capacity, increase muscle force, reduce dyspnea and improve quality of life and daily life activities in ILD patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of interstitial lung disease according to internationally established criteria
* Dyspnea on exertion
* Stable medical therapy
* Stable clinical condition at inclusion, with no infection or exacerbation in the previous 4 weeks

Exclusion Criteria:

* Co-morbidities that do not allow exercise training (unstable angina, recent myocardial infarction or cerebrovascular accident, active cancer, severe orthopedic disorders).
* Life expectancy below 3 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-04; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
changes in six minute walking distance after 6 months | 6 months
  primary outcome of rehabilitation programm

SECONDARY OUTCOMES:
Changes in dyspnea and quality of life scores (MMRC, CRDQ, SGRQ), | 3-6-12 months
Change in peripheral and respiratory muscle force | 3-6-12 months
Change in maximal exercise capacity | 3-6-12 months
Change in daily physical activity measured by Sensewear armband | 3-6-12 months
Changes in pulmonary function and blood gases at rest | 3-6-12 months
Change number of disease-related hospitalizations and survival | 3-6-12 months
Change in functional exercise capacity measured by the 6 minute walking distance | 12 months
To evaluate feasibility and safety of pulmonary rehabilitation in interstitial lung disease | 6 months
Changes in six minute walking distance | at 3, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Pérez-Bogerd, MD, Principal Investigator — KU Leuven; Wim Janssens, MD PhD, Principal Investigator — KU Leuven; Wim Wuyts, MD PhD, Principal Investigator — KU Leuven
Locations (1):
- Katholieke Universiteit Leuven, Leuven, Flanders, Belgium

REFERENCES:
- [Derived] Perez-Bogerd S, Wuyts W, Barbier V, Demeyer H, Van Muylem A, Janssens W, Troosters T. Short and long-term effects of pulmonary rehabilitation in interstitial lung diseases: a randomised controlled trial. Respir Res. 2018 Sep 20;19(1):182. doi: 10.1186/s12931-018-0884-y. PMID 30236104